CLINICAL TRIAL: NCT06780241
Title: Novel Characterization of Sex Specific Biologic Signatures in Valvular Heart Disease
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Deborah Kwon, MD, Principal Investigator, The Cleveland Clinic
Other Study IDs: 24-861
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Aortic Regurgitation; Mitral Regurgitation; Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Insufficiency; Mitral Valve Insufficiency; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: Cardiac MRI (CMR) with Magnetic Resonance Fingerprinting (MRF), fSENC (a new CMR technology which may detect subclinical signs of myocardial damage by measuring myocardial strain), Diffusion Tensor imaging (DTI), and chemical exchange transfer imaging with contrast at baseline and without contrast at follow up.
  Rapid Assessment of Physical Activity questionnaire Kansas City Cardiomyopathy Questionnaire
  Interventions: Diagnostic Test: CMR; Other: Quality of Life Questionnaire

INTERVENTIONS:
Diagnostic Test: CMR — CMR (with contrast at baseline and non-contrast at follow-up)
Other: Quality of Life Questionnaire — Rapid Assessment of Physical Activity questionnaire and the Kansas City Cardiomyopathy Questionnaire

SUMMARY:
This project aims to validate sex-specific biologic signatures associated with aortic valve disease developed in a large multicenter CMR registry, using unsupervised phenomapping.

The aim to use standard and advanced CMR techniques (MRF, DTI, chemical exchange transfer, and radiomics analysis) is to determine advanced CMR predictors of reverse remodeling following aortic valve surgery and develop sex-specific thresholds for risk. Infrastructure developed by this study will enable development of an innovative, scalable, sex-specific precision medicine cardiovascular imaging pipeline to determine overall risk and treatment response.

DETAILED DESCRIPTION:
Chronic valvular heart disease leads to significant left ventricular (LV) remodeling. Current national guidelines for surgical/procedural referral for valvular heart disease do not consider sex differences in presence of symptoms, LV remodeling and dysfunction. However, our prior research in patients with chronic aortic regurgitation, validated by our recent multicenter study, demonstrated that despite higher left ventricular function, and less ventricular dilation, females experienced more heart failure symptoms, fewer referrals for surgical intervention, and higher prevalence of adverse outcomes compared to males. Similarly, published HVTI data have demonstrated increased adverse outcomes in women referred for surgical mitral valve intervention.

Cardiac magnetic resonance (CMR) provides an exciting opportunity to characterize sex differences in LV remodeling.In combination with conventional CMR measures, novel CMR techniques such as Magnetic Resonance Fingerprinting (MRF), Diffusion Tensor imaging (DTI) and radiomics analysis provide tissue level specificity with potential to enhance phenomapping.

Limitations in understanding sex-specific remodeling patterns stem from heterogeneity of presentation, which confound traditional analytic methods. Phenomapping, a method of machine learning, clusters imaging features and patients into distinct phenotypic groups. Unsupervised phenomapping enables unbiased grouping of patients by both clinical characteristics as well as complex imaging features. In recent studies, this unbiased phenomapping approach demonstrates superior risk stratification of cardiac disease compared to traditional approaches that can be used to guide individualized treatment

The aim to use advanced CMR techniques (MRF, DTI, chemical exchange transfer, and radiomics analysis) is to determine advanced CMR predictors of reverse remodeling following procedural valve intervention and develop sex-specific thresholds for risk. Results from this study would enable the development of sex-specific precision medicine pathway, augmented by advanced imaging features, to better predict overall risk and treatment response, and thus enable novel patient selection criteria.

Study hypothesis: Radiomics, MRF, chemical exchange transfer, and DTI will elucidate distinct sex-specific biologic signatures, in addition to standard CMR imaging features, and are associated with adverse outcomes, and reverse remodeling following surgical/procedural valve intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90 years of age
* Suspected moderate or severe (2-3+ or more) aortic regurgitation, or moderate or more aortic stenosis on the basis of prior known clinical history, echocardiogram or cardiac MRI.

Exclusion Criteria:

* Acute traumatic cardiac injury
* Aortic dissection or aortic root rupture
* Congenital heart diseases such as patent ductus arteriosus, coarctation of aorta, ASD and VSD
* Presence of A-V fistula or intracardiac shunts
* Any contraindications to cardiac MRI including:

  * Patients with any MR-incompatible implant, including cardiac pacemakers or defibrillators, or older types of cerebral aneurysm clips.
  * Patients who weigh more than 440 lbs. or have a very wide waist circumference.
  * Patients with claustrophobia may have difficulty tolerating the exam.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with at least moderate Aortic Stenosis or Aortic Regurgitation who are scheduled for a surgical repair or replacement of their aortic valve.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in LV Dilation and/or change in LVEF | 6-12 months
  Significant change in LV remodeling will be defined as a change in EF by 10 units (reverse remodeling is defined at least 10 unit decrease) or change in LV end-diastolic/systolic volume by 10% (Reverse remodeling is defined as at least decrease in LV end-diastolic/systolic volume by 10%

SECONDARY OUTCOMES:
Change in Aortic Regurgiation | 6-12 months
  Change in Aortic Regurgitant Fraction will be modeled as a continuous variable, as well as a threshold change of 5 points or more, as measured by cardiac MRI
Change in BNP | 6-12 months
  NT-proBNP will be modeled as a continuous variable as well as a threshold change of 30% or decrease to level < 1000
Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) score | 6-12 months
  KCCQ will be modeled as a continuous variable, as well as a threshold change of 5 points or more.
  KCCQ scoring transforms Likert-scale answers into 0-100 scores (higher is better) for domains like Physical Limitation, Symptom Frequency, Quality of Life, and Social Limitations, with a summary score reflecting overall health, where 0-24 is very poor, 25-49 poor/fair, 50-74 fair/good, and 75-100 good/excellent health.
6 minute walk test | 6-12 months
  6 minute walk test will be modeled as a continuous variable as well as a threshold change of 30meters or more

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Kwon, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States